CLINICAL TRIAL: NCT03520842
Title: Study of Regorafenib in Combination With Oral Methotrexate for KRAS Mutated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Regorafenib and Methotrexate in Treating Participants With Recurrent or Metastatic KRAS Mutated Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heather Wakelee, Professor of Medicine (Oncology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-43398; NCI-2018-00413 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0097 (Other: OnCore)
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: KRAS Gene Mutation; Metastatic Malignant Neoplasm in the Brain; Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Methotrexate; merphos; Pharmacogenomic Variants; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (regorafenib, methotrexate) (Experimental): Participants receive regorafenib PO QD on days 1-21, and methotrexate PO twice weekly with 2-3 days apart on a 3 week on/ 1 week off cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Methotrexate; Other: Pharmacokinetic Study; Drug: Regorafenib

INTERVENTIONS:
Drug: Methotrexate — Given PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga

SUMMARY:
This phase II trial studies how well regorafenib works together with methotrexate in treating participants with metastatic non-squamous non-small cell lung cancer with tumors that harbor a KRAS mutation. Regorafenib is a targeted therapy that works on different cancer pathways to stop the growth of tumor cells and stop them from spreading. Methotrexate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving regorafenib and methotrexate together may work in treating participants with KRAS mutated non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression free survival (PFS) of the combination of regorafenib and methotrexate for metastatic KRAS mutated non-small cell lung cancer (NSCLC) patients who have received at least 1 prior systemic therapy.

SECONDARY OBJECTIVES:

I. To determine the objective response rate (ORR) of the combination of regorafenib and methotrexate for metastatic KRAS mutated NSCLC patients who have received at least 1 prior systemic therapy.

II. To determine the disease control rate (DCR) at 8 weeks of the combination of regorafenib and methotrexate for metastatic KRAS mutated NSCLC patients who have received at least 1 prior systemic therapy.

III. To determine the safety of the combination of regorafenib and methotrexate in metastatic KRAS mutated NSCLC patients who have received at least 1 prior systemic therapy, assessed as the number of subjects that experience a treatment-emergent adverse event.

IV. To determine the safety of the combination of regorafenib and methotrexate in metastatic KRAS-mutated NSCLC patients who have received at least 1 prior systemic therapy, assessed as the number (percent) of participants experiencing any dose-limiting toxicity (DLT).

V. To determine the pharmacokinetic parameters of methotrexate when combined with regorafenib (i.e., trough and maximum serum concentration [Cmax]).

OUTLINE:

Participants receive regorafenib orally (PO) once daily (QD) and methotrexate PO twice weekly with 2-3 days apart on a 3 week on / 1 week off schedule. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants will come in for an end of study treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmed diagnosis of non-squamous non-small cell lung cancer that is recurrent or metastatic.
* Documentation of pathogenic KRAS mutation
* Previous receipt of at least one systemic therapy for recurrent or metastatic disease OR previous receipt of adjuvant systemic therapy within 6 months of enrollment; there is no limit on number of prior therapies allowed
* Prior systemic therapy must be completed within 2 weeks of study treatment, with either improvement of clinically significant treatment-related toxicities to grade 0-1 OR stabilized to a new baseline
* Previously treated OR asymptomatic non-progressing < 1 cm untreated brain metastases are allowed
* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
* Ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) ≥ 1500/mm^3
* Platelet count ≥ 100,000 /mm^3
* Hemoglobin (Hb) ≥ 9 g/dL
* Serum creatinine ≤ 1.5x upper limit of normal (ULN) OR calculated (Cockcroft Gault formula) or measured creatinine clearance ≥ 50 mL/min for patients with creatinine levels > 1.5x ULN
* Total bilirubin ≤ 1.5x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x ULN (≤ 5x ULN for patients with liver involvement of their cancer)
* Must be able to swallow and retain oral medication
* Women patients of childbearing potential and men patients with women partners of childbearing potential must agree to use adequate contraception or agree to abstain from heterosexual activity beginning at the time of signing informed consent until at least 3 months after the last dose of study treatment; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not considered childbearing

Exclusion Criteria:

* Previously treated with regorafenib
* Known allergy to regorafenib or methotrexate
* Currently receiving another systemic standard or investigational anti-cancer therapy; prior investigational therapy must be completed within 4 half-lives (if known) or 2 weeks, whichever is longer; the maximal washout of investigational therapy will not exceed 4 weeks prior to study treatment; bone medications such as bisphosphonates and receptor activator of nuclear factor kappa-Β (RANK) ligand inhibitors permitted
* Leptomeningeal disease as documented by cerebrospinal fluid (CSF) cytology
* Clinically significant cardiovascular related disease including:

  * Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mmHg on repeated measurements, i.e., 3 or more separate days within one week) despite optimal medical management
  * Congestive heart failure - New York Heart Association (NYHA) class III or greater
  * Active coronary artery disease (i.e., unstable or new onset angina within 3 months of study treatment; myocardial infarction within 6 months of study treatment)
  * Clinically significant cardiac arrhythmias other than atrial flutter/fibrillation
  * Stroke, including transient ischemic attacks, within 6 months of study treatment
  * Other clinically significant arterial events, except for controlled asymptomatic pulmonary embolism, within 6 months of study treatment
* Clinically significant hemorrhage or bleeding event within 1 month of study treatment
* Uncontrolled symptomatic pleural effusion or ascites
* Known active additional malignancy that is undergoing or expected to undergo systemic treatment during duration of study participation
* Known history of human immunodeficiency virus (HIV) infection or known current active hepatitis B (i.e., hepatitis [Hep] B deoxyribonucleic acid [DNA] positive in prior 3 months) or hepatitis C infection (i.e., Hep C ribonucleic acid [RNA] positive in prior 3 months)
* Major surgical procedure (e.g., involving the opening of a major body cavity) within 4 weeks of study treatment; this does not apply to low risk procedures (i.e., thoracentesis; paracentesis; chest tube / PleurX catheter placement; line placement; needle biopsy of tumor; and bronchoscopy)
* Presence of a clinically significant non-healing wound, non-healing ulcer, or bone fracture
* Concomitant therapy required at time of first dose of study treatment, including:

  * Strong CYP3A4 inhibitors and CYP3A4 inducers
  * Regular use of nonsteroidal anti-inflammatory drugs (NSAIDs), proton pump inhibitors, and probenecid
* Women who are pregnant or breast feeding
* Any condition which, in the investigator's opinion, including substance abuse, medical, psychological or social conditions that makes the patient unsuitable for trial participation or may interfere with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Wakelee, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients signed consent, 18 were allocated to treatment.
Groups:
- Treatment (Regorafenib, Methotrexate): Participants receive regorafenib PO once daily (QD) on days 1-21, and methotrexate PO twice weekly with 2-3 days apart on a 3 week on/ 1 week off cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Regorafenib, Methotrexate)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Asian | 5
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Smoking Status [Count of Participants; unit: Participants]
  Never | 4
  Former | 14
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG: Eastern Cooperative Oncology Group
  The ECOG Performance Status scale indicates increasing levels of disability, with 0 indicating fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care; 3, capable of limited self-care; 4, completely disabled; and 5, dead.
  Participants
    0 | 2
    1 | 16
Disease Presentation [Count of Participants; unit: Participants]
  Recurrent | 11
  Metastatic | 7
History of Pleural Effusion [Count of Participants; unit: Participants]
  Yes | 9
  No | 9
Brain Metastases [Count of Participants; unit: Participants]
  Previously treated | 3
  Untreated stable | 1
  None | 14
Tumor Histology: Adenocarcinoma [Count of Participants; unit: Participants] | 18
KRAS Mutation Subtype [Count of Participants; unit: Participants]
  G12C | 5
  G12D | 6
  G12R | 2
  G12V | 2
  Q61L | 1
  G12C/K117N | 1
  G12S/A146V | 1
Previous Lines of Systemic Therapy [Count of Participants; unit: Participants]
  1 | 10
  2-3 | 5
  4-5 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS), measured from time of first study treatment until objective tumor progression as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria or death from any cause, whichever occurs earlier. PFS was calculated using the Kaplan-Meier method along with 95% confidence interval.
  RECIST v1.1 criteria are:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: From first study treatment assessed up to 15 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
months | 3.7 [1.8 to 8.6]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR; as determined by RECIST v1.1) will be assessed as the proportion (percent) of participants with either complete response (CR; disappearance of all target lesions) or partial response (PR; ≥ 30% decrease in the sum of the longest diameter of target lesions), with exact 95% confidence intervals based on a binomial distribution.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
percentage of participants | 16.7 [3.5 to 41.4]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) will be assessed as the proportion of complete responses (CR) + partial responses (PR) + stable disease (SD) after 8 weeks of treatment (+/- 1 week), as determined by using RECIST v1.1
Time Frame: At 8 weeks
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
percentage of participants | 66.7 [41.0 to 86.7]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Participants who experienced any treatment emergent adverse event and any ≥ grade 3 adverse event is reported.
Time Frame: Up to 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
Participants
  Any grade | 17
  ≥ grade 3 | 14

5. Secondary Outcome: Trough Serum Concentration of Methotrexate
Description: Pharmacokinetics (PK) of methotrexate when co-administered with regorafenib, as indicated by the trough serum concentration, was accessed by a fluorescent polarization immunoassay, and is reported as the mean with standard deviation. Participants treated with at least 1 dose of regorafenib and methotrexate and with at least one evaluable baseline pharmacokinetic sample and one follow up trough pharmacokinetic sample treated were included.
Time Frame: Cycle 1, Days 1, 8, 15, and 22
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
μmol/L
  Cycle 1, Day 1 | 0.04 (0.02)
  Cycle 1, Day 8 | 0.04 (0.01)
  Cycle 1, Day 15 | 0.05 (0.03)
  Cycle 1, Day 22 | 0.05 (0.02)

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of Methotrexate
Description: Pharmacokinetics (PK) of methotrexate when co-administered with regorafenib, as indicated by the maximum serum concentration (Cmax) of methotrexate, was assessed by a fluorescent polarization immunoassay, and is reported as the mean with standard deviation. Participants treated with at least 1 dose of regorafenib and methotrexate and with at least one evaluable Cmax pharmacokinetic sample were included in the assessment.
Time Frame: Cycle 1, Days 1, 8, and 15
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Treatment (Regorafenib, Methotrexate)
Number analyzed (Participants) | 18
μmol/L
  Cycle 1, Day 1 | 0.43 (0.23)
  Cycle 1, Day 8 | 0.60 (0.30)
  Cycle 1, Day 15 | 0.60 (0.43)

ADVERSE EVENTS:
Time Frame: Up to 38 months
Arm/Group | Treatment (Regorafenib, Methotrexate)
All-Cause Mortality (participants affected / at risk) | 2/18
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Regorafenib, Methotrexate) (N=18)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Thromboembolic event: pulmonary embolism (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Regorafenib, Methotrexate) (N=18)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Amylase increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Anemia (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Thrombocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Cardiomyopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Chills (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 3
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Esophageal stenosis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 9
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastroesphogeal reflux disease (Gastrointestinal disorders) | 2
Gas Pain (chest) (Gastrointestinal disorders) | 1
Hyperhidrosis (General disorders) | 1
Bleeding gums (General disorders) | 1
Headache (Nervous system disorders) | 3
Hiccups (Nervous system disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7
Hot flashes (Vascular disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Thyroid stimulating hormone increased (Investigations) | 1
Hyperbilirubinemia (Investigations) | 1
Lipase increased (Investigations) | 3
Localized edema (General disorders) | 3
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 9
Mucosal infection (Infections and infestations) | 1
Muscle cramp (bottom of feet) (Musculoskeletal and connective tissue disorders) | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Anosmia (Nervous system disorders) | 1
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 7
Palmar-plantar erthryodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Pancreatitis (Gastrointestinal disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Paresthesia (Nervous system disorders) | 2
Paronychia (Infections and infestations) | 1
Peripheral neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pulmonary hypertension (Vascular disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2
Urine output decreased (Renal and urinary disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Tenderness (Skin and subcutaneous tissue disorders) | 1
Finger fissures (Skin and subcutaneous tissue disorders) | 1
Scrotal erosion (Skin and subcutaneous tissue disorders) | 1
Papules (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Erythematous plaques (Skin and subcutaneous tissue disorders) | 1
Rash scalp (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (feet) (Skin and subcutaneous tissue disorders) | 1
scalp flaking (Skin and subcutaneous tissue disorders) | 1
pustule/cyst (labia) (Skin and subcutaneous tissue disorders) | 1
erythema (nasal region/scalp) (Skin and subcutaneous tissue disorders) | 1
skin peeling/blisters (fingers, feet, toes) (Skin and subcutaneous tissue disorders) | 1
Rash (face) (Skin and subcutaneous tissue disorders) | 1
Nonpruritic rash (upper chest, shoulders, back) (Skin and subcutaneous tissue disorders) | 1
Rash (groin) (Skin and subcutaneous tissue disorders) | 1
Sore throat (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 2
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03520842/Prot_SAP_000.pdf